CLINICAL TRIAL: NCT05230914
Title: Simple Imaging Versus Standard Imaging Selection in Stroke Patients for Endovascular Treatment: the NO-SELECT Randomized Trial
Brief Title: A Randomized Trial of Imaging Selection Modalities for Stroke Thrombectomy (NO-SELECT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: The First Affiliated Hospital of Hainan Medical University (Other Government); Dalian Central Hospital (Unknown); Huai'an First People's Hospital (Other)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NO-SELECT
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Ischemic; Stroke, Acute
Keywords: endovascular treatment; large vessel occlusion; acute ischemic stroke; computed tomography perfusion; non-contrast computed tomography; Alberta Stroke Program Early CT score
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple imaging (Experimental): NCCT and CTA will be used to screen patients for endovascular treatment
  Interventions: Other: Simplified imaging strategy
- Standard imaging (Active Comparator): NCCT-ASPECTS (pc-ASPECTS), CTA, and CTP will be used to screen patients for endovascular treatment
  Interventions: Other: Standard imaging strategy

INTERVENTIONS:
Other: Simplified imaging strategy — NCCT and CTA will be used to screen patients for endovascular treatment
  Arms: Simple imaging
Other: Standard imaging strategy — NCCT-ASPECTS (pc-ASPECTS), CTA, and CTP will be used to screen patients for endovascular treatment
  Arms: Standard imaging

SUMMARY:
Several studies suggest that advanced multi-modal imaging with CTP should be used to screen late time window stroke patients for thrombectomy. However, NCCT is more accessible when comparing with CTP. It is unclear whether the NCCT-based ASPECTS can be used as an imaging criterion to screen patients for thrombectomy.

The newly published MR CLEAN-LATE and TENSION trials used NCCT or CTA, but still relied on ASPECTS scores to evaluate and select patients for endovascular therapy. However, different trials have different time windows. The aim of this trial was to assess the clinical outcomes of stroke patients with anterior large vessel occlusion who selected by simple imaging (NCCT) comparing via standard imaging screening strategy (CTP/MRI). The hypothesis is that simple imaging is non-inferior to standard imaging selection strategy in terms of achieving favorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. The interval time from last known well to hospital arrival is within 24 hours;
3. Acute stroke confirmed by clinical symptoms or imaging examination;
4. Field Assessment Stroke Triage for Emergency Destination (FAST ED) ≥4;
5. Written informed consent is obtained from patients and/or their legal representatives.

Exclusion Criteria:

1. Allergy to radiographic contrast agents, or nitinol devices;
2. Currently pregnant or lactating (women patients);
3. Arterial tortuosity and/or other arterial disease that would prevent the device from reaching the target vessel;
4. Preexisting neurological or psychiatric disease that would confound the neurological functional evaluations;
5. Multiple vessel occlusion (e.g., bilateral anterior circulation, or occlusion of both anterior and posterior circulation);
6. Brain tumors with mass effect (except meningiomas) that are radiographically pleasant;
7. Intracranial aneurysm, arteriovenous malformation;
8. Any terminal illness with life expectancy less than 6 months;
9. Unlikely to be available for 90-day follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1846 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
favorable outcome at 90 days | 90 days post-endovascular treatment
  defined as modified Rankin scale score of 0 to 3. Modified Rankin scale score (mRS): scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.

SECONDARY OUTCOMES:
symptomatic intracranial hemorrhage within 48 hours | within 48 hours post-endovascular treatment
  symptomatic intracranial hemorrhage according to Heidelberg criteria
mortality at 90 days | 90 days post-endovascular treatment
  defined as the number of deaths observed divided by the number of subjects observed over the 90-day study period

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Xinqiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Wuyi Traditional Chinese Medicine Hospital, Jiangmen, Guangdong
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The 904th Hospital of CPLA, Wuxi, Jiangsu
  - Jingdezhen First People's Hospital, Jingdezhen, Jiangxi
  - Dalian Central Hospital, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: Yes
study data without patient information
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Related papers published 6 months later, the IPD will be shared
Access Criteria: yangqwmlys@163.com